CLINICAL TRIAL: NCT05118152
Title: Correlation Between 3D Echocardiography and Cardiopulmonary Exercise Testing in Patients With Single Ventricle: A Cross-sectional Observational Multicenter Prospective Study
Brief Title: Correlation Between 3D Echocardiography and Cardiopulmonary Exercise Testing in Patients With Single Ventricle
Acronym: VU3D
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0289
Record Dates: First submitted 2021-07-19; First posted 2021-11-11 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Single-ventricle; Congenital Heart Disease
Keywords: univentricular heart; Paediatric cardiology; cardiopulmonary exercise test; 3D echocardiography
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the leading cause of birth defects, with an incidence of 0.8%. Among CHD, univentricular heart disease or "single ventricle" is rare and complex. As a result of the improved patient care over the last decades, the number of children and adults with single ventricle is increasing significantly. Today, the main challenge is to ensure an optimal follow-up of these new patients in order to improve their life expenctancy as well as their quality of life (QoL). Currently, echocardiography and cardiopulmonary exercice test (CPET) are central in management of patients with single ventricle as part of good clinical practice guidelines.

Single ventricle volumes and function are very difficult to asses with conventional echocardiography because of their complex geometry. Indeed, single ventricle size and morphology vary depending on the patient characteristics and on the initial CHD (before surgical repair). That's why conventional 2D echocardiographic parameters are not reliable for single ventricle assessment.

Magnetic resonance imaging (MRI) is more effective in assessing single ventricle volumes and function. Nevertheless, MRI is not universally available, is not practical in many situations, is expensive, and is a relative contraindication in patients with pacemakers.

Over the past decade, the use of the 3D echocardiography has increased. This is an available tool that can assess ventricular function and volumes in few seconds. Recent studies shown a good correlation between 3D echocardiography and MRI for assessment of ventricular volumes and function in patient with CHD and especially in those with single ventricle.

Moreover, according to some authors, CPET parameters are strongly correlated with risk of hospitalization, risk of death, physical activity and quality of life, especially in patients with single ventricle.

To date, there is no study performed about the relationship between 3D echocardiography and CPET parameters in patients with single ventricle.

DETAILED DESCRIPTION:
This is a cross-sectional, observational, multicenter, and prospective study Eligible patients will be included during their usual medical check-up. As recommended by guidelines, patients with single ventricle have an 2D echocardiography and a CPET annualy. Data required for this study will be collected from patient medical record.

3D echography data acquisition will be performed using 2D ultrasound post-processing by TOMTEC software. No supplementary visit, directly related to the research, will be necessary. This study does not change the usual care management of the patient.

ELIGIBILITY:
Inclusion criteria:

* Patient over 8 years old with univentricular heart disease as defined by the ACC-CHD classification
* Agreement from adults or parents if minor patients
* CPET performed within the 6 months before or after performing echocardiography

Exclusion criteria:

* Cardiomyopathy unrelated to CHD (eg coronary artery disease, toxic cardiomyopathy)
* Significant clinical status change between performing CPET and performing echocardiography, according to the investigator's opinion

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a single ventricle or univentricular heart
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Association between single ventricle volumes and function parameters in 3D echocardiography | day 1
  Association between single ventricle volumes and function parameters in 3D echocardiography (End-diastolic volume, End-systolic volume, Stroke volume)

SECONDARY OUTCOMES:
Association between 3D echocardiography and clinical data collected | day 1
  Association between 3D echocardiography and clinical data collected in usual medical check-up.
Association between 3D echocardiography and quality of life data usually collected | day 1
  Association between 3D echocardiography and quality of life data usually collected.
ssociation between 3D echocardiography and 2D echocardiography data usually collected | day 1
  Association between 3D echocardiography and 2D echocardiography data usually collected.
Association between 3D echocardiography and blood test data usually collected. | day 1
  Association between 3D echocardiography and blood test data usually collected.
Association between 3D echocardiography and MRI data usually collected. | day 1
  Association between 3D echocardiography and MRI data usually collected.
Assessment of 3D echocardiography interobserver and intraobserver variability | day 1
  Assessment of 3D echocardiography interobserver and intraobserver variability.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER; Valentin FEMENIA, resident, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Femenia V, Pommier V, Huguet H, Iriart X, Picot MC, Bredy C, Lorca L, De La Villeon G, Guillaumont S, Pasquie JL, Matecki S, Roubertie F, Leobon B, Thambo JB, Jalal Z, Thomas J, Mouton JB, Avesani M, Amedro P. Correlation between three-dimensional echocardiography and cardiopulmonary fitness in patients with univentricular heart: A cross-sectional multicentre prospective study. Arch Cardiovasc Dis. 2023 Apr;116(4):202-209. doi: 10.1016/j.acvd.2023.02.002. Epub 2023 Mar 9. PMID 36966111